CLINICAL TRIAL: NCT04626713
Title: An Online Home-based Intervention for Anxiety Regulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Lee Tih Shih, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-220
Record Dates: First submitted 2020-10-05; First posted 2020-11-12 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Anxiety
Keywords: Anxiety; Biofeedback; Intervention
MeSH Terms: conditions — Anxiety Disorders | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will undergo a brief interactive psychoeducation session four times a week for two weeks. For each session, participants will wear a commercially available Electroencephalography (EEG) headset and play a downloaded online game for a total of 30 minutes. Participants can feel free to play the game for more than the instructed frequency during their 2-week intervention participation.
  Interventions: Device: Brain-Computer Interface
- Waitlist control (No Intervention): Participants in Waitlist Control will receive no intervention in the first four weeks of the study. After the Intervention group has completed treatment, participants in the Waitlist Control will then undergo the same intervention as the Intervention group.

INTERVENTIONS:
Device: Brain-Computer Interface — Brain-computer Interface (BCI) is a direct communication pathway between a human brain and an external device. Electroencephalography (EEG) is the best studied non-invasive interface facilitating such communication. Our technology will deliver a mindfulness-based anxiety regulation intervention through a neuro-/ bio-feedback-based game interface that is driven by an EEG algorithm.
  Arms: Intervention

SUMMARY:
The aim of this project is to evaluate the safety and acceptability of our online, home-based, personalized, neuro-technological mindfulness-based intervention in entraining anxiety regulation and ameliorating anxiety in healthy adults. Our technology will deliver a mindfulness-based anxiety regulation intervention through a neuro-/ bio-feedback-based game interface that is driven by an electroencephalography (EEG) algorithm. We hypothesize that the intervention would be safe and acceptable. In exploratory analyses, we further hypothesize that the intervention would help entrain anxiety regulation and ameliorate anxiety in healthy adults. Data will be analyzed quantitatively and qualitatively to inform development of our intervention and future research studies.

DETAILED DESCRIPTION:
Anxiety disorders, defined by excess worry, hyperarousal and fear, are amongst the most common class of psychiatric conditions in adults. Large population-based studies on anxiety disorders estimated a lifetime prevalence of 33.7% and a 12-month prevalence between 2.4% and 29.8%. In Singapore, however, studies have only established the prevalence of a limited range or anxiety disorders. In a nationwide, cross-sectional, epidemiological survey, the lifetime prevalence of anxiety disorders, specifically Generalized Anxiety Disorder and Obsessive-Compulsive Disorder, rose from 0.9% and 3.0% respectively in 2010, to 1.6% and 3.6% in 2016. If untreated, anxiety disorders could result in a range of personal and societal costs, such as interpersonal dysfunctions, employment, physical health, social functioning, and frequent primary and acute care visits, resulting in a poor quality of life.

A large proportion of the population experiences subclinical symptoms of anxiety disorders which impede daily functioning and well-being, but most often do not seek professional help or fall below the radar of psychiatric services. Current treatment guidelines recommend pharmacotherapy (i.e. selective serotonin reuptake inhibitors [SSRIs] or venlafaxine) and psychotherapy (i.e. cognitive behavior therapy [CBT]) as first-line treatments for anxiety disorders. Unfortunately, SSRIs are associated with an increased risk of suicide in young adults. Thus, local practices often incorporate more psychological therapies in the treatment of anxiety disorders. However, CBT is labor-intensive and time-consuming - which is incompatible with the demanding lifestyle Singaporeans lead these days. Moreover, therapeutic outcomes are also very much therapist dependent. Due to the fear of stigma that is particularly salient in the local context, individuals with anxiety may be deterred from engaging with therapists. Even if these individuals do receive adequate treatment, existing literature shows that outcomes for recommended treatment modalities are sub-optimal at best, i.e. overall mean remission rate of CBT is 51% while pharmacotherapy is significantly lower. With the low rates of help-seeking behaviors and dismal success rates of existing therapies, novel interventions for anxiety are apposite and vital.

The benefits of mindfulness-based interventions have been extensively researched in anxiety disorders in recent years. Improvements reported across a range of outcomes include enhanced ability to cope with stress, reduced depressive and anxiety symptom severity, as well as improved sleep quality, all of which lead to increased life satisfaction and overall well-being. Not all anxiety regulation strategies are helpful, and mindful emotion regulation presents one promising strategy by cultivating a changing of relationship with one's emotions. Specifically, this strategy facilitates reduced reactivity to emotional stimuli by encouraging one to meet, accept, and detach from one's aversive feelings, thoughts, and ineffective habitual responses. Unfortunately, clinically anxious individuals with no experience in such practices could find it challenging to engage in them as they often require a high degree of individual discipline. Coupled with the fact that sustained practice is crucial to yield the benefits of mindfulness practice, an appealing mode of treatment delivery is necessary. To this end, gamification strategies could be useful: gamification strategies have been shown useful in motivating health-related behaviors through interaction with the immersive interventional programs. Recent preliminary studies have also suggested that neuro-/ biofeedback-based relaxation and mindfulness training is useful for both healthy and anxious individuals.

Accordingly, we have developed an online, home-based, personalized, neuro-technological mindfulness-based intervention and seek to conduct a preliminary study with healthy young adults to evaluate its safety and acceptability. Our technology will deliver a mindfulness-based anxiety regulation intervention through a neuro-/ bio-feedback-based game interface that is driven by an electroencephalography (EEG) algorithm. We hypothesize that the intervention would be safe and acceptable. We further hypothesize that the intervention would help entrain anxiety regulation and ameliorate anxiety in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 and 35 years old (inclusive).
* Literate in English.
* Computer literate and has access to a Windows 10 desktop or laptop
* Beck Anxiety Inventory II total score ≥ 16

Exclusion Criteria:

* Diagnosis (as defined by DSM-5) of: any anxiety disorder induced by medication, substance, or another medical condition; obsessive compulsive disorder; bipolar disorder; any psychotic disorder (lifetime); intellectual disability (i.e. IQ < 70); autism spectrum disorder; attention-deficit/ hyperactivity disorder
* History of substance or drug use disorder (as per DSM-5 criteria) within the last 3 months
* Neurological disorders or insults (e.g. epilepsy, cerebrovascular accidents)
* Metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites
* Gross visual and hearing impairments
* Irregular heart rhythms or heart problems, severe visual or hearing impairment
* Prior experience with mindfulness-based therapy (e.g. mindfulness-based stress reduction [MBSR], mindfulness-based cognitive therapy [MBCT])

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Inventory II (BAI-II) | Intervention group: Changes from baseline anxiety symptoms (week 1) to post-intervention (week 4) and follow-up (week 7). Waitlist control group: Changes from baseline anxiety symptoms (week 1) to pre-intervention (week 4) and post-intervention (week 7).
  21-item questionnaire being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
State-trait Anxiety Inventory (STAI) | Intervention group: Changes from baseline anxiety symptoms (week 1) to post-intervention (week 4) and follow-up (week 7). Waitlist control group: Changes from baseline anxiety symptoms (week 1) to pre-intervention (week 4) and post-intervention (week 7).
  4-point Likert scale and consisting of 40 questions measuring two types of anxiety - state and trait anxiety.
Usability questionnaire (System usability questionnaire) | Intervention group: Week 4 (post-intervention).
  Participants will rate their agreeableness on 10 statements regarding their satisfaction and ease of use of the training components on a 5-point Likert scale. Participants will also answer three qualitative questions regarding their satisfaction and ease of use.
IT Anxiety Scale (ITAS) | Intervention group: Week 4 (post-intervention).
  7-point Likert scale and consisting of 12 statements measuring participants' anxiety towards information and communication technologies.
Usability questionnaire (System usability questionnaire) | Waitlist control group: Week 7 (post-intervention).
  Participants will rate their agreeableness on 10 statements regarding their satisfaction and ease of use of the training components on a 5-point Likert scale. Participants will also answer three qualitative questions regarding their satisfaction and ease of use.
IT Anxiety Scale (ITAS) | Waitlist control group: Week 7 (post-intervention).
  7-point Likert scale and consisting of 12 statements measuring participants' anxiety towards information and communication technologies.
Number of Adverse Events/Serious Adverse Events Reported | Throughout the intervention period (2 weeks), which are weeks 2 and 3 for the intervention group.
  The total number and severity rating of all adverse events reported will be collated at the end of the study.
Number of Adverse Events/Serious Adverse Events Reported | Throughout the intervention period (2 weeks), which are weeks 5 and 6 for the waitlist control group.
  The total number and severity rating of all adverse events reported will be collated at the end of the study.

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | Intervention group: Changes from baseline sleep quality (week 1) to post-intervention (week 4) and follow-up (week 7). Waitlist control group: Changes from baseline sleep quality (week 1) to pre-intervention (week 4) and post-intervention (week 7).
  19-item questionnaire assessing sleep quality over a 1-month time interval.
Insomnia Severity Index (ISI) | Intervention group: Changes from baseline insomnia symptoms (week 1) to post-intervention (week 4) and follow-up (week 7). Waitlist control group: Changes from baseline (week 1) to pre-intervention (week 4) and post-intervention (week 7).
  7-item instrument assessing the severity of both nighttime and daytime components of insomnia.
Difficulties in Emotion Regulation Scale (DERS-SF) | Intervention group: Changes from baseline emotional regulation (week 1) to post-intervention (week 4) and follow-up (week 7). Waitlist control group: Changes from baseline (week 1) to pre-intervention (week 4) and post-intervention (week 7).
  18-item measure used to identify emotional regulation issues in adults.
Mindfulness Awareness Attention Scale (MAAS) | Intervention group: Changes from baseline mindfulness (week 1) to post-intervention (week 4) and follow-up (week 7). Waitlist control group: Changes from baseline mindfulness (week 1) to pre-intervention (week 4) and post-intervention (week 7).
  15-item questionnaire assessing individual differences in the frequency of mindful states over time.
Depression Anxiety Stress Scale (DASS-21) | Intervention group: Changes from baseline depression, anxiety and stress (week 1) to post-intervention (week 4) and follow-up (week 7). Waitlist control group: Changes from baseline (week 1) to pre-intervention (week 4) and post-intervention (week 7).
  21-item questionnaire measures the severity of symptoms of depression, anxiety and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Tih Shih Lee, MD PHD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore